CLINICAL TRIAL: NCT00558116
Title: Treating Carpal Tunnel Syndrome With Dynamic Splinting: A Randomized, Controlled, Trial
Brief Title: Treatment of Carpal Tunnel Syndrome With Dynamic Splinting
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Advanced Centers for Orthopaedic Surgery and Sports Medicine (Other)
Collaborators: Dynasplint Systems, Inc. (Industry)
Responsible Party: Stacey H Berner, MD, Advanced Centers for Orthopaedic Surgery and Sports Medicine
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 101010
Record Dates: First submitted 2007-11-12; First posted 2007-11-14 (Estimated); Last update posted 2008-05-13 (Estimated); Status verified 2008-05

CONDITIONS: Carpal Tunnel Syndrome
Keywords: Carpal Tunnel Syndrome; Dynamic Splinting; Nerve Conduction Studies; Splinting; Levine Katz Survey
MeSH Terms: conditions — Carpal Tunnel Syndrome | interventions — Splints

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Treatment with Dynasplint device
  Interventions: Device: Dynamic splinting
- 2 (No Intervention): Control group; does not receive conservative or surgical treatment.
  Interventions: Device: Dynamic splinting

INTERVENTIONS:
Device: Dynamic splinting — The Dynasplint carpal tunnel device will be worn for 30 minutes, twice daily, for 60 consecutive days.

SUMMARY:
The Purpose of this study is to examine the effect of using the Carpal Tunnel Dynasplint® System on patients diagnosed with CTS in a randomized, controlled, cross-over study.

DETAILED DESCRIPTION:
This study will compare the efficacy of treating Carpal tunnel Syndrome with the Dynasplint® Systems device as compared to a non-treatment control group utilizing a randomized, controlled, cross-over study design. The dependant variables in this study are each patient's score on a Levine-Katz disability and pain scale test, and the change in nerve conduction of the median nerve that was tested upon diagnosis. The independent variables will include three different patient groups separated by randomization. The first group of subjects (selected randomly) will be fit with a therapeutic, functional Carpal Tunnel Dynasplint® versus the second, control patients will not be treated with dynamic splinting for the first sixty (60) days. After the initial sixty (60) days, the original control patients will be fit with a functional Carpal Tunnel Dynasplint® system and this will allow examiner to evaluate for further variance between subject groups, allowing the third group to be a Cross-Over group.

The METHODS for this multi-centered study include recruiting patients from multiple hand surgeons and neurologists and these patients will have been diagnosed with following the physicians' physical examination and a nerve conduction test of the median nerve. The subjects then will be briefed on this study and sign an informed consent as required by the IRB before participating. Subjects who do consent will then be given the Levine-Katz disability and pain scale test, and prior to being fit with the Carpal Tunnel Dynasplint® Subjects will be taught how to use a Carpal Tunnel Dynasplint® properly and after being fit with the Carpal Tunnel Dynasplint® each subject will be required to complete a weekly report showing compliance to the wearing and treatment schedule, and they must attend regular, monthly examinations by the referring physician. After the initial sixty (60) days in the study each subject will repeat the three lead conduction test of the median nerve.

Control subjects at this point will be fit with the Carpal Tunnel Dynasplint® systems becoming Cross-Over subjects and their final nerve conduction test will be administered after they have worn the Carpal Tunnel Dynasplint® system for sixty (60) days. Upon discharge from this study all subjects will also retake the Levine-Katz disability and pain scale test.

Eighty (80) SUBJECTS will be recruited following diagnosis of CTS (using nerve conduction testing of the median nerve for differential diagnosis) and group assignment will be determined through randomization following each patient's completion of the informed consent required by the IRB. All patients randomly selected to start in the experimental group will be fit with functional Carpal Tunnel Dynasplint® and the control group subjects will not be fit until after sixty (60) days. When they are ultimately fit, they will then be categorized as "Cross-Over" subjects to measure continued variance between all groups.

The DURATION for patients enrolled in this study will be sixty (60) days for the experimental subjects and the control subjects will spend their first sixty (60) days as a control role without treatment. However, following sixty days the initial control subjects but then they will be refit with a functional Carpal Tunnel Dynasplint® as a "Cross-Over" subject for an additional sixty (60) days, which makes the control subjects duration in this study 120 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients must exhibit one of the following symptoms of CTS: numbness, tingling, or pain in the wrist or hand
* Patients will be ≥18 years old and of either gender
* Patients will agree and be able to sign a voluntary consent to participate form
* Nerve Conduction study results as follows:

Sensory conduction latency to peak greater than 3.7ms when measured with ring pick up on the volar surface of the index finger measured 14cm from stimulation across the wrist at the median nerve Motor conduction latency to take off greater than 4.2ms when measured with disc pick up on the abductor pollicis brevis muscle measured 8 cm from stimulation across the wrist at the median nerve

-

Exclusion Criteria:

* Patients that have thenar atrophy of the hand
* Patients that are currently undergoing manual, hand therapy
* Patients that have been previously diagnosed with cervical radiculopathy
* Patients whose examination shows evidence of a "Double Crush" syndrome
* Pregnancy
* Nerve Conduction study results as follows:

Sensory conduction latency to peak less than 3.7ms when measured with ring pick up on the volar surface of the index finger measured 14cm from stimulation across the wrist at the median nerve Motor conduction latency to take off less than 4.2ms when measured with disc pick up on the abductor pollicis brevis muscle measured 8cm from stimulation across the wrist at the median nerve

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2007-05; Primary Completion 2008-11 (Estimated); Study Completion 2008-12 (Estimated)

PRIMARY OUTCOMES:
Change in Nerve Conduction Test results | 60 days

SECONDARY OUTCOMES:
Change in score of Levine-Katz outcome survey | 60 days

CONTACTS AND LOCATIONS:
Overall Officials: Stacey H Berner, MD, Principal Investigator — Advanced Centers for Orthopaedic Surgery and Sports Medicine
Locations (1):
- Advanced Centers for Orthopaedic Surgery and Sports Medicine, Owings Mills, Maryland, United States